CLINICAL TRIAL: NCT04011228
Title: Sex-specific Relationship of Epigenetics Based Modifications in the Saliva and Blood With the Occurence of Type 2 Diabetes
Brief Title: Epigenetics Based Diagnosis of Diabetes in Saliva and Blood Samples
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Alexandra Kautzky-Willer, Principal Investigator, Medical University of Vienna
Other Study IDs: EPI-1090
Record Dates: First submitted 2019-03-13; First posted 2019-07-08 (Actual); Last update posted 2019-09-03 (Actual); Status verified 2019-08

CONDITIONS: Prediabetic State; Diabetes Mellitus, Type 2; Ectopic Lipids; Epigenetics Based Modifications
MeSH Terms: conditions — Prediabetic State; Diabetes Mellitus, Type 2 | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Type 2 diabetic patients
  Interventions: Diagnostic Test: Blood sampling; Diagnostic Test: Saliva and blood samples; Diagnostic Test: Magnet Resonance Spectroscopy
- Prediabetic patients
  Interventions: Diagnostic Test: Blood sampling; Diagnostic Test: Saliva and blood samples; Diagnostic Test: Magnet Resonance Spectroscopy
- Women with gestational diabetes
  Interventions: Diagnostic Test: Blood sampling; Diagnostic Test: Saliva and blood samples; Diagnostic Test: Magnet Resonance Spectroscopy
- Healthy control subjects
  Interventions: Diagnostic Test: Blood sampling; Diagnostic Test: Saliva and blood samples; Diagnostic Test: Magnet Resonance Spectroscopy
- Pregnant women without gestational diabetes
  Interventions: Diagnostic Test: Blood sampling; Diagnostic Test: Saliva and blood samples; Diagnostic Test: Magnet Resonance Spectroscopy

INTERVENTIONS:
Diagnostic Test: Blood sampling — After a fasting period over night blood samples will be taken.
Diagnostic Test: Saliva and blood samples — After a fasting period over night blood and saliva samples will be taken for the investigation of epigenetics based modifications.
Diagnostic Test: Magnet Resonance Spectroscopy — The amount of ectopic lipids in the liver, heart and the skeletal muscle will be measured using 1H-magnetic resonance spectroscopy.

SUMMARY:
The aim of the present study is to investigate epigenetics based modifications and biomarkers in the saliva and blood in diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetic patients
* prediabetic patients
* women with gestational diabetes
* healthy control subjects without diabetes
* healthy pregnant women

Exclusion Criteria:

* cancer disease
* infectious diseases such as hepatitis or HIV
* malignoms
* patients with claustrophoby

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: In the present study prediabetic patients, type 2 diabetic patients, women with gestational diabetes and healthy control subjects will be included.
Sampling Method: Non-Probability Sample
Enrollment: 224 (Estimated)
Dates: Start 2016-02-29 (Actual); Primary Completion 2019-12-11 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
Specifying the microRNAs in saliva in diabetic patients | 1 hour
  Characterization of microRNAs in saliva of prediabetic and type 2 diabetic patients, as well as in women with gestational diabetes and healthy control subjects.

SECONDARY OUTCOMES:
Correlation of the percentage of liver fat with miRNA´s in diabetic patients. | 1 hours
  Correlation of miRNA´s in the saliva with the amount of intrahepatic liver fat.
Correlation of the percentage of heart fat with miRNA´s in diabetic patients | 1 hour
  Correlation of miRNA´s in the saliva with the amount of ectopic lipids in the heart.
Correlation of the percentage of the content of fat in the skeletal muscle with miRNA´s in diabetic patients. | 1 hour
  Correlation of miRNA´s in the saliva with the amount of ectopic lipids in the skeletal muscle.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Kautzky-Willer, Univ.Prof.Dr., Principal Investigator — Department of Internal Medicine III, Clinical Division of Endocrinology and Metabolism, Unit of Gender Medicine, Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Derived] Klepochova R, Leutner M, Bastian M, Krebs M, Weber M, Trattnig S, Kautzky-Willer A, Krssak M. Muscle-Specific Relation of Acetylcarnitine and Intramyocellular Lipids to Chronic Hyperglycemia: A Pilot 3-T 1H MRS Study. Obesity (Silver Spring). 2020 Aug;28(8):1405-1411. doi: 10.1002/oby.22846. PMID 32820618